CLINICAL TRIAL: NCT05174923
Title: An Observational Study to Assess the Feasibility and Variability of Physical Assessments Performed by People 45 Years of Age or Older Who Are Overweight or Obese
Brief Title: Variability of Physical Assessments in an Older Population That is Overweight or Obese
Status: Completed | Type: Observational
Sponsor: Versanis Bio, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VER201-OBS-032
Record Dates: First submitted 2021-11-05; First posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Obesity; Aging
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Age Range 45 to </= 60
  Interventions: Behavioral: Short Performance Physical Battery (SPPB Test); Behavioral: 30 Second Chair Stand Test (30CST); Behavioral: Hand grip dynamometry
- Age Range 61 to </= 75
  Interventions: Behavioral: Short Performance Physical Battery (SPPB Test); Behavioral: 30 Second Chair Stand Test (30CST); Behavioral: Hand grip dynamometry
- Age >/= 76
  Interventions: Behavioral: Short Performance Physical Battery (SPPB Test); Behavioral: 30 Second Chair Stand Test (30CST); Behavioral: Hand grip dynamometry

INTERVENTIONS:
Behavioral: Short Performance Physical Battery (SPPB Test) — The SPPB includes balance stands, a 4-meter walk and 5 timed chair stands.
Behavioral: 30 Second Chair Stand Test (30CST) — The 30CST measures the number of times a person can rise from a seated to standing position within 30 seconds.
Behavioral: Hand grip dynamometry — Grip strength is used as a marker of overall muscle strength.

SUMMARY:
Variability of physical assessments in an older population that is overweight or obese.

DETAILED DESCRIPTION:
The purpose of this study is to understand difficulty in obtaining physical assessment measurements and assess the variability of these assessments when performed by people who are overweight or obese. Data collected in this protocol will be used to inform the design of future clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* A written informed consent must be obtained before any study-related assessment is conducted.
* Men and women aged ≥ 45.
* BMI ≥ 30 or BMI ≥ 27 with one or more obesity-associated comorbidities (e.g. hypertension, cardiovascular disease, hyperlipidemia, elevated fasting blood sugar levels, sleep apnea).
* Participants must be able to communicate well with the Investigator and comply with the study requirements.

Exclusion Criteria:

* Participant weight > 150 kg.
* Systolic blood pressure < 90 or > 180 or diastolic blood pressure <50 or >100.
* Heart rate ≤ 50 or ≥ 100.
* Unstable medical condition that would put the participant at risk by performing the study assessments.
* Chronic medical condition rendering participants unable to perform the assessment, e.g., severe knee osteoarthritis.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 60 male and female participants 45 years of age or older who are overweight or obese will be enrolled. To ensure data are collected from a wide age range, 20 participants will be enrolled per specified age ranges. The study population must include at least 40% females in the overall study.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
To assess the variability of Short Physical Performance Battery (SPPB, scored from 0-12) results within and between participants. | Baseline (+7 day window)
To assess the variability of the 30 Second Chair Stand (30CST) results within and between participants. | Baseline (+7 day window)
To assess the variability of grip strength results (kg) with the use of a hand grip dynamometer within and between participants. | Baseline (+7 day window)
To assess the variability of the individual Short Physical Performance Battery (SPPB) with subsets (subsets of Balance, Gait and Chair Stand scored 0-4) within participants. | Baseline (+7 day window)
To compare the variability between the 5 Repetition Sit to Stand (5STS) subtest of the SPPB and 30CST. | Baseline (+7 day window)
To assess the correlation between bioelectrical impedance analysis (BIA) and waist circumference (WC) as well as body mass index (BMI). | Baseline (+7 day window)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - CNS Healthcare, Jacksonville, Florida
  - CNS Healthcare, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No